CLINICAL TRIAL: NCT03064763
Title: A Phase 1, Multi-center, Open-Label, Dose De-escalation Study to Evaluate the Safety and Efficacy of Talimogene Laherparepvec in Japanese Subjects With Unresectable Stage IIIB-IV Malignant Melanoma
Brief Title: Study to Evaluate the Safety/ Efficacy of T-VEC in Japanese Subjects With Unresectable Stage IIIB-IV Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20140270
Record Dates: First submitted 2017-02-09; First posted 2017-02-27 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Unresectable Stage IIIB-IV Malignant Melanoma
Keywords: Unresectable Stage IIIB-IV Malignant Melanoma
MeSH Terms: interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Talimogene laherparepvec (Experimental): Participants will receive talimogene laherparepvec administered by intralesional injection only into injectable cutaneous, subcutaneous, and nodal tumors, with or without image ultrasound guidance.
  On Day 1 (Week 0), the initial dose of talimogene laherparepvec will be up to 4.0 mL of 10^6 Plaque forming units per millilitre (PFU/mL). Subsequent doses of talimogene laherparepvec will be up to 4.0 mL of 10^8 or 10^7 PFU/mL. The second dose is to be administered 3 weeks (+ 5 days) after the initial dose, and subsequent doses were to be given every 2 weeks (+ 3 days).
  Interventions: Drug: Talimogene laherparepvec

INTERVENTIONS:
Drug: Talimogene laherparepvec — Talimogene laherparepvec will be administered as an intralesional injection.
  Other Names: Imlygic; T-VEC

SUMMARY:
There are 2 fold of purposes for this study. 1 is to evaluate safety and tolerability and the other is to study the anti-tumor effects of talimogene laherparepvec in Japanese participants with unresectable stage IIIB-IV malignant melanoma.

DETAILED DESCRIPTION:
This is a phase 1, multicenter, open-label study of talimogene laherparepvec in Japanese participants with unresectable stage IIIB-IVM1c malignant melanoma that are candidates for intralesional therapy. The Screening period is 28 days prior to study enrollment. There will be a Treatment period, Safety Follow-up period and a Long Term Follow-up period.

The Screening Period: Informed consent will be obtained prior to screening procedures. Screening procedures to determine eligibility include: medical history (including concomitant medications, prior therapy for melanoma and BRAF status (if known)), physical exam, vital signs, assessment of Eastern Cooperative Oncology Group (ECOG) performance level status, electrocardiogram (ECG), laboratory assessments (including hepatitis serology), baseline tumor assessments, and adverse events assessment.

Treatment Period: Initially, 6 Dose Limiting Toxicity (DLT)-evaluable participants will be enrolled and treated at 100% dose regimen of talimogene laherparepvec (Up to 4.0 mL of 10_6 PFU/mL followed by a dose of up to 4.0 mL of 10_8 PFU/mL). Upon demonstration of safety based on DLT incidence in the first 6 participants, an additional 12 participants will be enrolled and treated at Dose 1 to obtain additional safety data. If dose de-escalation is needed based on the DLT evaluation of first 6 participants, then additional 6 participants will be treated at lower dose (up to 4.0 mL of 10_6 PFU/mL followed by a dose of up to 4.0 mL of 10_7PFU/mL). The duration of treatment will vary for each participants. Participants will be treated until the participant has a DLT during the DLT evaluation period, participant has achieved a Complete Response, no injectable lesions, clinically relevant (resulting in clinical deterioration or requiring change in therapy) disease progression beyond 24-weeks of treatment, or safety concern, whichever occurs first. Maximum treatment duration will be 48 months. The total study duration for an individual participant can be up to 4 years.

Drug Administration: If the participants are found to be eligible to take part in this study, they will receive talimogene laherparepvec by intralesional injection only into injectable cutaneous, subcutaneous, and nodal tumors, with or without image ultrasound guidance. The first injection of talimogene laherparepvec will take place on day 1 (week 0). The second injection should be administered 3 weeks (+ 5 days) after the initial injection. Subsequent injections should be given every 2 weeks (± 3 days).

Study Visits: The participant will have a physical exam along with vital signs and ECOG. At any study visit blood may be collected to monitor health and safety, and effects of talimogene laherparepvec. Adverse events and medications taken will be reviewed at each study visit. The tumor assessment, physical exams, and ECOG performance status will be completed after 12 (± 1) weeks on treatment (ie, day 1 of week 11), and then every 12 (± 1) weeks (eg, weeks 23, 35, 47 etc.), or more frequently if clinically indicated, until Progressive disease beyond 6 months of treatment or until the start of a new anticancer therapy.

Central Lab tests: Blood for herpes simplex virus type-1 (HSV-1) Antibody Serostatus will collected within 3 days prior to dose at day 1 (week 0) and at week 5. Throughout the trial any participant developing a lesion of suspected herpetic origin will have a swab of the lesion for presence of talimogene laherparepvec DNA obtained within 3 days of the event.

Exposure to talimogene laherparepvec by the healthcare providers of the participant and/or close contacts will be assessed.

Safety Follow Visit: A safety follow-up visit will be performed 30 (+7) days after the last dose. The participant will have a physical exam, have vital signs taken, assessment of ECOG status and have weight measured. Adverse events will be assessed as well as the concomitant medications. Routine bloodwork and tumor response assessments will be performed.

Long-Term Follow-up Visits: Follow-up for survival status and, if applicable, commencement of any subsequent anticancer melanoma therapy will occur every 12 weeks (± 28 days) by phone or clinic visit for all participants who permanently discontinue talimogene laherparepvec for any reason other than withdrawal of full consent for up to 24 months after the last participant is enrolled in the study. For participants that discontinue talimogene laherparepvec for reason other than disease progression, the following additional procedures will be conducted during the long-term follow-up: radiographic tumor imaging, clinical tumor assessments, ECOG Performance Status assessments, reporting of pregnancy or lactation, assessment of swabs of lesions of suspected herpetic origin for presence of talimogene laherparepvec DNA, and tumor response assessments until documented disease progression beyond 24-weeks of treatment, until the start of a new anticancer therapy, or end of study, whichever is earliest. If a participant discontinues therapy more than 24 months after the last participant was enrolled in the study, when the long-term follow-up period ends, they will not enter long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of melanoma
* Participants with stage IIIB to IVM1c melanoma that is not surgically resectable
* Participant who is treatment naive and is determined by the physician to be not suitable or eligible for the approved systemic anticancer drug therapy in Japan. Participant may also have received prior systemic anticancer treatment consisting of chemotherapy, immunotherapy, or targeted therapy. Treatment for melanoma must have been completed at least 28 days prior to enrollment.
* Candidate for intralesional therapy (ie, disease is appropriate for direct injection or through the use of ultrasound guidance, where appropriate) defined as one or more of the following:

  * at least 1 injectable cutaneous, subcutaneous, or nodal melanoma lesion greater or equal to 10 mm in longest diameter, OR
  * multiple injectable melanoma lesions that in aggregate have a longest diameter of greater or equal to 10 mm
* Measurable disease defined as one or more of the following:

  * at least 1 melanoma lesion that can be accurately and serially measured in at least 2 dimensions and for which the greatest diameter is greater or equal to 10 mm as measured by contrast-enhanced or spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or ultrasound for nodal/soft tissue disease (including lymph nodes)
  * at least 1 greater or equal to 10 mm longest diameter superficial cutaneous or subcutaneous melanoma lesion as measured by calipers
  * multiple superficial melanoma lesions which in aggregate have a total diameter of greater or equal to 10 mm
* Serum lactate dehydrogenase (LDH) levels less than or equal to 1.5 X upper limit of normal (ULN) within 28 days prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Other Inclusion Criteria May Apply.

Exclusion Criteria:

* Clinically active cerebral metastases. Participants with up to 3 cerebral metastases may be enrolled, provided that all lesions have been adequately treated with stereotactic radiation therapy (including Gamma Knife) or craniotomy, with no evidence of progression and have not required steroids for at least 2 months prior to enrollment.
* Greater than 3 visceral metastases (this does not include lung metastases or nodal metastases associated with visceral organs). For participants with less than or equal to 3 visceral metastases, no lesion greater than 3 cm in longest dimension and liver lesions must be stable for at least 1 month prior to enrollment.
* Bone metastases
* Primary ocular or mucosal melanoma
* History or evidence of symptomatic autoimmune disease (eg, pneumonitis, glomerulonephritis, vasculitis, or other), or history of autoimmune disease that required systemic treatment (ie, use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past 2 months prior to enrollment.
* Active herpetic skin lesions or prior complications of herpetic infection (eg, herpetic keratitis or encephalitis).
* Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use.
* Previous treatment with talimogene laherparepvec
* Other investigational procedures while participating in this study are excluded.
* Known to have acute or chronic active hepatitis B infection, acute or chronic active hepatitis C infection or human immunodeficiency virus (HIV) infection
* Participant has known sensitivity to bovine- or porcine derived components or to any of the products or components to be administered during dosing.
* History of other malignancy within the past 3 years
* Other Exclusion Criteria May Apply

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (9):
- Japan (9):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Shinshu University Hospital, Matsumoto-shi, Nagano
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Osaka International Cancer Institute, Osaka, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Yamazaki N, Isei T, Kiyohara Y, Koga H, Kojima T, Takenouchi T, Yokota K, Namikawa K, Yi M, Keegan A, Fukushima S. A phase I study of the safety and efficacy of talimogene laherparepvec in Japanese patients with advanced melanoma. Cancer Sci. 2022 Aug;113(8):2798-2806. doi: 10.1111/cas.15450. Epub 2022 Jun 30. PMID 35656636
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 18 participants were enrolled at 8 centers in Japan from March 2017 until January 2023.
Groups:
- Talimogene Laherparepvec: Participants received talimogene laherparepvec administered by intralesional injection only into injectable cutaneous, subcutaneous, and nodal tumors, with or without image ultrasound guidance.
  On Day 1 (Week 0), the initial dose of talimogene laherparepvec was up to 4.0 mL of 10^6 Plaque forming units per millilitre (PFU/mL). Subsequent doses of talimogene laherparepvec were up to 4.0 mL of 10^8 or 10^7 PFU/mL. The second dose was administered 3 weeks (+ 5 days) after the initial dose, and subsequent doses were given every 2 weeks (+ 3 days). Participants could receive talimogene laherparepvec for a maximum treatment duration of 48 months.
Period: Overall Study
Arm/Group | Talimogene Laherparepvec
Started | 18
Received Treatment | 18
Completed | 9
Not Completed | 9
Not completed — Lost to Follow-up | 1
Not completed — Death | 8

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of talimogene laherparepvec.
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced One or More Dose Limiting Toxicities (DLTs)
Description: DLTs were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4
  Events were considered DLTs, if judged by the investigator to be related to study treatment:
  Grade 4 non-hematologic toxicity Grade 3 non-hematologic toxicity lasting > 3 days despite optimal supportive care (grade 3 fatigue not a DLT)
  Grade 3 or higher non-hematologic laboratory value reported as an adverse event if:
  medical intervention is required, or abnormality leads to hospitalization, or abnormality persists for > 1 week (Laboratory values that persist for > 1 week but are deemed not clinically important per both investigator and sponsor were not considered DLTs) Febrile neutropenia grade 3 or 4 Thrombocytopenia < 25 x 10^9/L associated with bleeding event requiring intervention Serious herpetic event (eg, herpetic encephalitis, encephalomyelitis, or disseminated herpetic infection) Grade 5 toxicity Any other intolerable toxicity leading to permanent discontinuation of study treatment
Time Frame: Day 1 to Day 35
Population: The DLT Analysis Set: all participants who had the opportunity to be followed for at least 35 days on treatment from the initial dosing (unless discontinued due to DLT) and received at least 1 dose of talimogene laherparepvec.
Measure: Count of Participants; unit: Participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 18
Participants | 0

2. Primary Outcome: Durable Response Rate (DRR) Using Modified World Health Organization (WHO) Response Criteria
Description: DRR using WHO response criteria was defined as the percentage of participants who experienced objective response (complete response [CR] or partial response [PR]) lasting continuously for ≥ 6 months that starting any time within 12 months of initiating treatment.
  CR: Complete disappearance of all index lesions, including any new tumors which might have appeared.
  PR: Achieving a 50% or greater reduction in the SPD of the perpendicular diameters of all index lesions at the time of assessment as compared to the sum of the products of the perpendicular diameters of all index lesions at baseline (Day 1).
Time Frame: Day 1 up to the maximum time on treatment or follow-up at primary data cutoff date (03 August 2020): 89.1 weeks of treatment and 37 months of follow-up
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of talimogene laherparepvec.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 18
Percentage of participants | 11.1 [1.4 to 34.7]

3. Secondary Outcome: Overall Response Rate (ORR) Using Modified World Health Organization (WHO) Response Criteria
Description: ORR was defined as the percentage of participants who experienced an objective response of CR or PR per modified WHO response criteria among the set of participants analyzed.
Time Frame: Day 1 to end of study, maximum time to end of study was 212.6 weeks
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of talimogene laherparepvec.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 18
Percentage of participants | 11.1 [1.4 to 34.7]

4. Secondary Outcome: Time to Response (TTR) Using Modified World Health Organization (WHO) Response Criteria
Description: TTR was defined as the time from the first treatment administration to the first incidence of a confirmed CR or PR according to modified WHO response criteria among the set of participants analyzed.
  TTR was estimated using Kaplan-Meier (KM) method.
Time Frame: Day 1 to end of study, maximum time to end of study was 212.6 weeks
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of talimogene laherparepvec.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 18
Months | NA [8.08 to NA] — The median TTR or upper limit could not be estimated due to insufficient number of participants who experienced either CR or PR.

5. Secondary Outcome: Duration of Response (DOR) Using Using Modified World Health Organization (WHO) Response Criteria
Description: DOR was defined as the time from the date of an initial response (CR or PR) to the earlier of progressive disease (PD) or death. Participants who had not ended their response at the time of analysis were censored at their last evaluable tumor assessment.
  PD: A > 25% increase in the sum of the products of the perpendicular diameters of all index tumors since baseline, or the unequivocal appearance of a new tumor since the last response assessment time point.
  DOR was estimated using Kaplan-Meier (KM) method.
Time Frame: Day 1 to end of study, maximum time to end of study was 212.6 weeks
Population: Responders among Safety Analysis Set: all enrolled participants who received at least 1 dose of talimogene laherparepvec who experienced a response of either CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 2
Months | NA [11.07 to NA] — The median DOR or upper limit could not be estimated due to insufficient number of participants who experienced either CR or PR.

6. Secondary Outcome: Progression Free Survival (PFS) Using Using Modified World Health Organization (WHO) Response Criteria
Description: PFS was defined as the interval from the first dose to the earlier of PD per modified WHO response criteria or death from any cause; otherwise, PFS was censored at the last evaluable tumor assessment.
  PFS was estimated using Kaplan-Meier (KM) method.
Time Frame: Day 1 to end of study, maximum time to end of study was 212.6 weeks
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of talimogene laherparepvec.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 18
Months | 3.07 [2.56 to 5.78]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the interval from first dose to the event of death from any cause; otherwise, OS was censored at the date the participant was last known to be alive.
  OS was estimated using Kaplan-Meier (KM) method.
Time Frame: Day 1 to end of study, maximum time to end of study was 212.6 weeks
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of talimogene laherparepvec.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 18
Months | NA [17.51 to NA] — The median OS or upper limit could not be estimated due to insufficient number of participants who experienced death.

ADVERSE EVENTS:
Time Frame: Deaths: From enrollment to end of study, up to maximum of 212.6 weeks; SAE and non-serious AEs: Day 1 (post 1st dose) to 30 days after last dose. Median (min, max) duration of treatment overall was 23.14 (3.1, 201.6) weeks
Arm/Group | Talimogene Laherparepvec
All-Cause Mortality (participants affected / at risk) | 8/18
Serious Adverse Events (participants affected / at risk) | 6/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (N=18)
Malaise (General disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Enteritis infectious (Infections and infestations) | 1
Epiglottitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (N=18)
Anaemia (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 2
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 2
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 9
Jaundice cholestatic (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Bacterial infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 5
Subcutaneous abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Vitiligo (Skin and subcutaneous tissue disorders) | 1
Contrast media allergy (Immune system disorders) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03064763/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT03064763/SAP_001.pdf